CLINICAL TRIAL: NCT07093268
Title: A Phase 1 Study to Determine the Safety and Tolerability of Continuous Intrathecal Riluzole in Patients With Progressive Ambulatory Amyotrophic Lateral Sclerosis
Brief Title: Safety of Intrathecal Riluzole in Patients With Amyotrophic Lateral Sclerosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brain Trust Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITR2023
Record Dates: First submitted 2024-05-08; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: Neurodegenerative Diseases; Nervous System Diseases; Neuromuscular Diseases
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neurodegenerative Diseases; Nervous System Diseases; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: Open label, competitive recruitment.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Intrathecal riluzole continuous infusion up to 0.2 mg / hr.
  Interventions: Drug: Intrathecal Riluzole

INTERVENTIONS:
Drug: Intrathecal Riluzole — Intrathecal infusion of riluzole for 6 weeks followed by 6 months treatment with safety committee approval.

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of intrathecal riluzole in adults with amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
ALS/MND is a progressive motor neurone disease. Oral riluzole is approved for the treatment of ALS/MND in Australia as well as other countries. Unfortunately, in pill form, the drug's efficacy is limited by erratic absorption from the gut, dosing is limited by liver toxicity, and patients often experience brain fog as a troubling side effect. Evidence from dogs suggests that receiving the same drug through an implanted pump that infuses it directly into the cerebrospinal fluid around the cells that support breathing, allows these cells to get 3 to 10 times as much riluzole , and guarantees that it is always there at the desired amount. In addition, this delivery approach should not contribute to increased brain fog.

Patients who have demonstrated the ability to tolerate oral riluzole will have a SynchroMed® II Infusion Pump and Ascenda ® Intrathecal Catheter implanted. Once deemed medically appropriate, 6-weeks of continuous IT riluzole will be administered. Safety and tolerability will be assessed by a safety committee for the first 3 participants enrolled. With Safety Committee approval, these participants will continue on 6-months of treatment and a further 7 participants will be enrolled for a total of 32 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older.
* Participants are ambulatory with or without an assistive device.
* Sporadic or familial ALS diagnosis with possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria.
* Slow vital capacity (SVC) measure ≥70% of predicted for gender, height, and age.
* Medically able to undergo implantation of the SynchroMed II Infusion Pump according to the judgment of the investigator, or the presence of a previously implanted IT pump (not to be used for concurrent IT infusion of another IT agent).
* Capable of reading and providing informed consent and following study procedures.
* Geographic accessibility to the study center and the ability to travel to the clinic for study visits by ground transportation.
* Women must not be able to become pregnant (eg, post menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and 3 months after study completion. Adequate contraception includes: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal (patch or contraceptive ring, for example) contraception), intrauterine device in place for ≥3 months, barrier method in conjunction with spermicide, or another adequate method.
* Taking and tolerating oral riluzole 50 mg twice a day for at least 30 days prior screening and willingness to continue oral riluzole throughout duration of the study.
* Patients may take other drugs approved for treatment of ALS at the dose prescribed by their neurologist.

Exclusion Criteria:

* Participants with bulbar-onset ALS
* Participants at risk of increased bleeding or uncontrolled bleeding during the SynchroMed II Infusion Pump implantation or following explant. This includes but is not limited to:

  1. Anatomical factors at or near the site of implantation;
  2. Underlying disorders of the coagulation cascade or platelet function (eg, hemophilia, Von Willebrand's disease, liver disease);
  3. Administration of antiplatelet or anticoagulant medication within 7 days before or after pump implantation (eg, aspirin, clopidogrel bisulfate, rivaroxaban, nonsteroidal anti-inflammatory agents [NSAIDs]), or
  4. Use of nutritional supplements (eg, St John's Wort) within 7 days before or after pump implantation.
* Presence of infection including but not limited to: meningitis, ventriculitis, skin infection, bacteremia, or septicemia.
* Testing positive for HIV (anti-HIV antibody), HBV (HBV surface antigen) or HCV (anti-HCV antibody; HCV RNA if anti-HCV antibody is positive) at screening.
* Inability to have the infusion pump implanted ≤ 2.5 cm below the skin surface.
* Body weight and size unable to accept the infusion pump bulk and weight.
* Spinal anomalies which would complicate the implantation and fixation of the catheter for IP delivery.
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) value > 2.0 times the upper normal.
* A life expectancy of less than 6 months, based on the judgment of the investigator.
* Presence of tracheostomy.
* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair the ability of the participant to provide informed consent, per investigator judgment.
* History of active substance abuse within the prior year.
* At risk for committing suicide per investigator judgment.
* Clinically significant history of unstable or severe cardiac, oncologic, hepatic, or renal disease, or other medically significant illness.
* Pregnant women or women currently breastfeeding.
* Exposure to any investigational drug, device, or biologic within 30 days of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with abnormal vital signs | 6 weeks
  Serial assessment of adverse events, vital signs (blood pressure, pulse, respiratory rate and temp)
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with with abnormal physical examination findings | 6 weeks
  Serial assessment of abnormal findings in a neurological examination for ALS patients
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with abnormal neurological exam findings | 6 weeks
  Serial assessment all adverse events, neurological examination
Safety and tolerability of 0.2mg/hr intrathecal, infusion of intrathecal riluzole, Number of participants with with abnormal laboratory tests results | 6 weeks
  Serial assessment all abnormal findings in clinical laboratory test results
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with abnormal findings in the Neuropathic Pain Scale (NPS) | 6 weeks
  Serial assessment all abnormal findings in the Neuropathic Pain Scale (NPS)
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with adverse events, Columbia-Suicide Severity Rating Scale (C-SSRS). | 6 weeks
  Serial assessment all adverse events in the Columbia-Suicide Severity Rating Scale (C-SSRS).

SECONDARY OUTCOMES:
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with abnormal vital signs | 6 months
  Serial assessment of adverse events, vital signs (blood pressure, pulse, respiratory rate and temp)
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with abnormal physical examination findings | 6 months
  Serial assessment of abnormal findings in a neurological examination for ALS patients
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with abnormal neurological exam findings | 6 months
  Serial assessment all adverse events, neurological examination
Safety and tolerability of 0.2mg/hr intrathecal, infusion of intrathecal riluzole, Number of participants with with abnormal laboratory tests results | 6 months
  Serial assessment all abnormal clinical laboratory test results
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with abnormal findings in the Neuropathic Pain Scale (NPS) | 6 months
  Serial assessment all abnormal findings in the Neuropathic Pain Scale (NPS)
Safety and tolerability of 0.2mg/hr intrathecal infusion of intrathecal riluzole, Number of participants with adverse events, Columbia-Suicide Severity Rating Scale (C-SSRS). | 6 months
  Serial assessment all adverse events in the Columbia-Suicide Severity Rating Scale (C-SSRS).

OTHER OUTCOMES:
Exploratory - Measure of changes in blood and cerebrospinal fluid biomarkers and urinary p75 | 9 months
  Measure of BDNF, pNFH and NfL) and cerebrospinal fluid (pNFH, NfL, Chit-1, CHI3L1, MCP-1, IL-6, IL-8, IL-17, IL-18, MIP-1α, TNF-α, CRP, 8-oxodG, Ferritin, BDNF, NGF, p75ECD biomarkers
Exploratory - Measure of clinical outcome of Handheld dynamometry (HHD) during dosing and post treatment periods. | 9 months
  Measure of Handheld dynamometry (HHD)
Exploratory - Tracheostomy free survival | 9 months
  To compare tracheostomy free survival for all participants with data from historical controls
Exploratory - Measure of clinical outcome measures during dosing and post treatment periods. | 9 months
  Measure of the ALS Functional Rating Scale - Revised (ALSFRS-R),
Exploratory - Measure of clinical outcome measures during dosing and post treatment periods. | 9 months
  Measure of slow vital capacity (SVC),
Exploratory - Measure of clinical outcome measures during dosing and post treatment periods. | 9 months
  Measure of the Rasch-Built Overall ALS Disability Scale (ROADS),
Exploratory - Measure of clinical outcome measures during dosing and post treatment periods. | 9 months
  Measure of the Amyotrophic Lateral Sclerosis-Specific Quality of Life-short form (ALSSQOL-SF)

CONTACTS AND LOCATIONS:
Overall Officials: David Schultz, Dr, Principal Investigator — Flinders Medical Centre; Antony Winkel, Dr, Principal Investigator — Sunshine Coast University Hospital
Locations (2):
- Australia (2):
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia

IPD SHARING:
Plan to Share IPD: No